CLINICAL TRIAL: NCT06449768
Title: Effectiveness Of Suprachoroidal Injection In Diabetic Macular Edema
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSRSW/Batch-Fall22/719
Record Dates: First submitted 2024-05-25; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Diabetic Macular Edema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Diabetic Macular Edema — observing the eye behavior in Diabetic Macular Edema

SUMMARY:
It will investigate a novel treatment approach for diabetic macular edema (DME), which causes vision impairment in diabetic patients. It will focuse on the efficacy and safety of administering triamcinolone acetonide via suprachoroidal injection, targeting the space between the sclera and choroid.

DETAILED DESCRIPTION:
This method aims to enhance drug delivery to the retina, potentially improving outcomes compared to conventional treatments. Participants receive suprachoroidal injections, and the study measures changes in macular thickness and visual acuity. The study's findings could offer a promising alternative to existing DME treatments, aiming to provide better management of the condition and improved patient quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Above 30 years old patients male and female
* Diabetic patient
* Diabetic patient for more than 2 years
* Macular thickness of more than 280um

Exclusion Criteria:

* Patient below 30 years
* Patients having media opacity
* Patients with other systemic problems
* Uncooperative patients

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic Macular Edema patient having Diabetes for more than 2 years
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-10-28 (Estimated)

PRIMARY OUTCOMES:
Visual Acuity Testing | 12 Months
  Visual acuity testing evaluates the participants' ability to discern letters or symbols at a standardized distance, providing a measure of vision clarity. This tool helps determine the functional improvement in vision.
Optical Coherence Tomography | 12 months
  OCT is employed to assess changes in macular thickness, providing detailed cross-sectional images of the retina. This non-invasive imaging technique helps quantify the extent of macular edema and monitoring

CONTACTS AND LOCATIONS:
Locations (1):
- Lions Medical Complex , Main Market, Gulberg ll, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No